CLINICAL TRIAL: NCT01876485
Title: Point-of-care Health Literacy and Activation Information to Improve Diabetes Care
Acronym: EPIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CRE 12-426
Record Dates: First submitted 2013-06-10; First posted 2013-06-12 (Estimated); Results first posted 2019-06-19 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-03

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; health literacy; patient activation; goals of care
MeSH Terms: conditions — Diabetes Mellitus; Patient Participation | interventions — Long-Term Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: Empowering Patients in Chronic Care (EPIC) (Experimental): Patients in the intervention arm will receive the Empowering Patients in Chronic Care group training sessions consisting of 6 one-hour group sessions occurring over a 6-month period. Group sessions will consist of behavioral coaching focused on diabetes management. Following each group-session, patients enrolled in the intervention arm will meet with a designated member of their primary care team to personalize diabetes goals and action plans.
  Interventions: Behavioral: Empowering Patients in Chronic Care (EPIC)
- Arm 2: Enhanced Usual Care (EUC) (Active Comparator): The Enhanced Usual Care (EUC) arm will serve as a concurrent control group to compare to the intervention arm of the study. Patients randomized to EUC will be referred to the PACT RN Care Manager for diabetes management, and will also receive a packet of educational materials regarding diabetes management, including a letter delineating the diabetes management resources available at their facility.
  Interventions: Behavioral: Enhanced Usual Care (EUC)

INTERVENTIONS:
Behavioral: Empowering Patients in Chronic Care (EPIC) — EPIC group training sessions consisting of 6 one-hour group sessions occurring over a 6-month period. Group sessions will consist of behavioral coaching focused on diabetes management. Following each group-session, patients enrolled in the intervention arm will meet with a designated member of their primary care team to personalize diabetes goals and action plans.
  Arms: Arm 1: Empowering Patients in Chronic Care (EPIC)
Behavioral: Enhanced Usual Care (EUC) — Patients randomized to EUC will be referred to the PACT RN Care Manager for diabetes management, and will also receive a packet of educational materials regarding diabetes management, including a letter delineating the diabetes management resources available at their facility.
  Arms: Arm 2: Enhanced Usual Care (EUC)

SUMMARY:
This hybrid effectiveness/implementation trial will be conducted in two phases over four years. In Phase 1, the investigators will evaluate the process of implementing a collaborative, diabetes goal-setting intervention (Empowering Patients in Chronic Care [EPIC]) personalized to self-reported patient activation and functional health literacy (FHL) levels into routine primary care practices. In Phase 2, the investigators will conduct a randomized, clinical trial to compare the effectiveness of EPIC to enhanced usual care (EUC). In Phase 2, the investigators will conduct a randomized clinical trial enrolling 284 Veterans with poorly controlled diabetes defined by average hemoglobin A1c over the last six months of >= 8% to receive EPIC or enhanced usual care (EUC). Consented subjects will be allocated evenly between EPIC and EUC. EPIC consists of six 1-hour group sessions focusing on 1) Your Health, Your Values, 2) Diabetes ABCs, 3) Setting Goals and Making Action Plans, 4) Communication with Your Health Care Provider, 5) Staying Committed to Your Goals, and 6) Reviewing and Planning for the Future. After each group session, a one-on-one session between a designated PACT member and patient participants will focus on collaborative goal-setting. Patients randomized to EUC will be referred to the PACT RN Care Manager for diabetes management, and will also receive a packet of educational materials regarding diabetes management, including a letter delineating the diabetes management resources available at their facility. Study measurements using self-reported questionnaires and blood tests to assess blood sugar control will be obtained at baseline, post-intervention, and post-six month maintenance period.

DETAILED DESCRIPTION:
Project Background: Diabetes mellitus is a highly prevalent chronic condition, affecting one in four Veterans who use the Veterans Affairs (VA) health care system. Self-management skills are critical for controlling diabetes and reducing its cardiovascular sequela. Providing diabetic patients with effective self-management training and support can be challenging due to time constraints at primary care encounters and limited clinician training with behavior change. The investigators have previously demonstrated that a group-based, VA primary care intervention to help patients set highly effective, evidence-based diabetes goals had a positive impact on both diabetes self-efficacy and hemoglobin (Hb) A1c levels. This study aims to evaluate the process of implementing a collaborative goal-setting intervention personalized to patient activation and health literacy levels (i.e. Empowering Patients in Chronic Care [EPIC]) into routine PACT care and to evaluate the effectiveness of this intervention relative to usual care.

Project Objectives: Specific Aim 1: Assess effective processes for and costs associated with implementing a collaborative diabetes goal-setting intervention personalized to patient activation and FHL (i.e., EPIC) into the routine workflows of PACTs. H1: Formative measures within the PARIHS framework (evidence, context, facilitation) will be associated with implementation of EPIC (defined by reach, adoption, cost effectiveness, and fidelity measures) into routine PACT care. Specific Aim 2: Evaluate the effectiveness of delivering collaborative goal-setting personalized to patient activation and FHL on clinical (HbA1c) and patient-centered (Diabetes Distress Scale) outcomes among eligible patients in enrolled PACTs. H2: Patients receiving collaborative goal-setting personalized to activation and FHL levels will have significant improvements in a) HbA1c and b) Diabetes Distress Scale levels, respectively, at post-intervention compared with patients receiving enhanced usual care. H3: Patients receiving collaborative goal-setting personalized to activation and FHL levels will maintain significant improvements in a) HbA1c and b) Diabetes Distress Scale levels at post-maintenance follow-up, respectively, compared with patients receiving enhanced usual care.

Project Methods: In Phase 1 of the study, the investigators will implement EPIC into routine PACT care. The investigators will conduct a mixed-methods formative evaluation that includes 33-48 key informant interviews with VA leadership, clinicians, and staff and an assessment of organizational readiness for change. This evaluation will identify how group and one-on-one sessions of EPIC can best be implemented into routine workflows of PACT. In Phase 2, the investigators will conduct a randomized clinical trial enrolling 284 patients with poorly controlled diabetes defined by average hemoglobin A1c of 8% to receive EPIC or enhanced usual care. The patient will serve as the unit of randomization. EPIC consists of six 1-hour group sessions focusing on 1) Your Health, Your Values, 2) Diabetes ABCs, 3) Setting Goals and Making Action Plans, 4) Communication with Your Health Care Provider, 5) Staying Committed to Your Goals, and 6) Reviewing and Planning for the Future. After each group session, a one-on-one session between a designated PACT member and patient participants will focus on collaborative goal-setting. Designated PACT members will be trained to personalize goal-setting using patient-reported activation and health literacy data. The investigators will collect laboratory and survey data at baseline, post-intervention, and post-maintenance phase. The investigators will evaluate the effectiveness of personalized goal-setting compared to enhanced usual care on clinical (e.g., hemoglobin A1c) and patient-centered (e.g., Diabetes Distress Scale) outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Veterans receiving primary care at VA study sites who are enrolled in the panels of participating primary care teams
* Veterans with ICD-9-CM and/or ICD-10 codes indicating a diagnosis of diabetes
* Veterans with an average HbA1c level > 8% in the prior 6 months

Exclusion Criteria:

The investigators will exclude Veterans with the following clinical conditions that would render participation in a group clinic inappropriate:

* metastatic cancer or receiving hospice care
* limited life expectancy
* clinician recommendations to not titrate therapy due to prior history of significant hypoglycemic events
* age <18 years
* active bipolar or psychotic disorder

The investigators will also exclude Veterans, who at the time of screening:

* cannot attend monthly group clinic sessions due to transportation or availability barriers
* have significant cognitive impairment
* have active substance-abuse disorders
* are not comfortable discussing their health and health care in a peer-group setting Patients will be secondarily excluded if their HbA1C level falls below 7.5% at baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2015-07-13 (Actual); Primary Completion 2018-02-09 (Actual); Study Completion 2018-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: LeChauncy D. Woodard, MD MPH, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (3):
- United States (3):
  - Jesse Brown VA Medical Center, Chicago, IL, Chicago, Illinois
  - Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Arney J, Thurman K, Jones L, Kiefer L, Hundt NE, Naik AD, Woodard LD. Qualitative findings on building a partnered approach to implementation of a group-based diabetes intervention in VA primary care. BMJ Open. 2018 Jan 21;8(1):e018093. doi: 10.1136/bmjopen-2017-018093. PMID 29358425
- [Result] Woodard LD, Adepoju OE, Amspoker AB, Virani SS, Ramsey DJ, Petersen LA, Jones LA, Kiefer L, Mehta P, Naik AD. Impact of Patient-Centered Medical Home Implementation on Diabetes Control in the Veterans Health Administration. J Gen Intern Med. 2018 Aug;33(8):1276-1282. doi: 10.1007/s11606-018-4386-x. Epub 2018 Apr 2. PMID 29611089
- [Derived] Banks J, Amspoker AB, Vaughan EM, Woodard L, Naik AD. Ascertainment of Minimal Clinically Important Differences in the Diabetes Distress Scale-17: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2023 Nov 1;6(11):e2342950. doi: 10.1001/jamanetworkopen.2023.42950. PMID 37966840
- [Derived] Woodard L, Amspoker AB, Hundt NE, Gordon HS, Hertz B, Odom E, Utech A, Razjouyan J, Rajan SS, Kamdar N, Lindo J, Kiefer L, Mehta P, Naik AD. Comparison of Collaborative Goal Setting With Enhanced Education for Managing Diabetes-Associated Distress and Hemoglobin A1c Levels: A Randomized Clinical Trial. JAMA Netw Open. 2022 May 2;5(5):e229975. doi: 10.1001/jamanetworkopen.2022.9975. PMID 35507345

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 2: Enhanced Usual Care (EUC): The Enhanced Usual Care (EUC) arm will serve as a concurrent control group to compare to the intervention arm of the study. Patients randomized to EUC will be referred to the Patient Aligned Care Team (PACT) Registered Nurse (RN) Care Manager for diabetes management, and will also receive a packet of educational materials regarding diabetes management, including a letter delineating the diabetes management resources available at their facility.
  Enhanced Usual Care (EUC): Patients randomized to EUC will be referred to the PACT RN Care Manager for diabetes management, and will also receive a packet of educational materials regarding diabetes management, including a letter delineating the diabetes management resources available at their facility.
Period: Overall Study
Arm/Group | Arm 1: Empowering Patients in Chronic Care (EPIC) | Arm 2: Enhanced Usual Care (EUC)
Started | 140 | 140
Post-Intervention (4 months after baseline) | 125 | 129
Maintenance (10 months after baseline) | 116 | 114
Completed | 116 | 114
Not Completed | 24 | 26

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Empowering Patients in Chronic Care (EPIC) | Arm 2: Enhanced Usual Care (EUC) | Total
Number analyzed (Participants) | 140 | 140 | 280
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 49 | 95
  >=65 years | 94 | 91 | 185
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.39 (8.57) | 66.94 (8.34) | 67.17 (8.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 131 | 133 | 264
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 11 | 33
  Not Hispanic or Latino | 116 | 125 | 241
  Unknown or Not Reported | 2 | 4 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 140 | 140 | 280
Percent Glycosylated Hemoglobin (HbA1c) [Mean (Standard Deviation); unit: Percent/DCCT] | 9.11 (1.60) | 9.06 (1.32) | 9.08 (1.46)
Diabetes Distress Scale (DDS) [Mean (Standard Deviation); unit: Units on a scale] | 2.41 (1.05) | 2.45 (1.02) | 2.43 (1.03)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Percent Glycosylated Hemoglobin (HbA1c) Levels During Intervention
Description: Measures of HbA1c will be taken to assess average blood glucose levels throughout the study as an indicator of diabetes control.
Time Frame: HbA1c levels will be measured at baseline, four months, and ten months.
Population: Although not all of the 140 per group with HbA1c at baseline completed each the post-intervention and maintenance assessments, intent to treat analyses were conducted which enabled us to use the full 140 across time points.
Measure: Mean (Standard Deviation); unit: Percentage/DCCT
Arm/Group | Arm 1: Empowering Patients in Chronic Care (EPIC) | Arm 2: Enhanced Usual Care (EUC)
Number analyzed (Participants) | 140 | 140
Percentage/DCCT
  Baseline | 9.11 (1.60) | 9.06 (1.32)
  4 Months: number analyzed (Participants) | 125 | 125
  4 Months | 8.61 (1.27) | 9.04 (1.70)
  10 Months: number analyzed (Participants) | 116 | 110
  10 Months | 8.68 (1.53) | 8.79 (1.55)
Statistical Analysis 1: Comparison: Arm 1: Empowering Patients in Chronic Care (EPIC) vs Arm 2: Enhanced Usual Care (EUC); We compared group differences in HbA1c at 4. The value of HbA1c at 4 months was the dependent variable, treatment group was the independent variable, and baseline HbA1c was a covariate. Power calculations were based on effect sizes for the HbA1c in similar trial that revealed small-to-medium effect sizes. Our goal was to include 130 patients in each arm. The randomized samples (n = 140 EPIC, n = 140 EUC) exceed the required 130 per group; Test type: Superiority; p = 0.003, proc mixed in SAS (multilevel modeling); Numerator degrees of freedom = 1 for both models (4mo and 10mo) and denominator degrees of freedom vary based on multiple imputation; Mean Difference (Final Values) = 0.43
Statistical Analysis 2: Comparison: Arm 1: Empowering Patients in Chronic Care (EPIC) vs Arm 2: Enhanced Usual Care (EUC); We compared group differences in HbA1c at 10 months. The value of HbA1c at 10 months was the dependent variable, treatment group was the independent variable, and baseline HbA1c was a covariate. Power calculations were based on effect sizes for the HbA1c in similar trial that revealed small-to-medium effect sizes. Our goal was to include 130 patients in each arm. The randomized samples (n = 140 EPIC, n = 140 EUC) exceed the required 130 per group; Test type: Superiority; p = .60, proc mixed in SAS (multilevel modeling); [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = .11

2. Primary Outcome: Change in Diabetes Specific Quality of Life
Description: The Diabetes Distress Scale (DDS) will be used to assess diabetes quality of life throughout the study. Minimum value: 1; Maximum value: 6. Higher scores indicate a higher level of diabetes distress.
Time Frame: Diabetes specific quality of life will be measured at baseline, four months, and ten months.
Population: Seven participants did not complete the DDS at baseline. Therefore, sample sizes for DDS are lower than for HbA1c.
  Although not all of the 138/135 per group with DDS at baseline completed each the post-intervention and maintenance assessments, intent to treat analyses were conducted which enabled us to use the full number across time points.
Measure: Mean (Standard Deviation); unit: Units On A Scale
Arm/Group | Arm 1: Empowering Patients in Chronic Care (EPIC) | Arm 2: Enhanced Usual Care (EUC)
Number analyzed (Participants) | 138 | 135
Units On A Scale
  Baseline | 2.41 (1.05) | 2.45 (1.02)
  4 Months: number analyzed (Participants) | 123 | 126
  4 Months | 2.02 (0.81) | 2.30 (0.99)
  10 Months: number analyzed (Participants) | 114 | 111
  10 Months | 1.96 (0.76) | 2.27 (1.05)
Statistical Analysis 1: Comparison: Arm 1: Empowering Patients in Chronic Care (EPIC) vs Arm 2: Enhanced Usual Care (EUC); We compared group differences in DDS at 4 months. The value of DDS at 4 months was the dependent variable, treatment group was the independent variable, and baseline DDS was a covariate. Power calculations were based on effect sizes for the DDS in similar trial that revealed small-to-medium effect sizes. Our goal was to include 130 patients in each arm. The randomized samples (n=138 EPIC, n=135 EUC) exceed the required 130 per group; Test type: Superiority; p = 0.003, proc mixed in SAS (multilevel modeling); Mean Difference (Final Values) = 0.30
Statistical Analysis 2: Comparison: Arm 1: Empowering Patients in Chronic Care (EPIC) vs Arm 2: Enhanced Usual Care (EUC); We compared group differences in DDS at 10 months. The value of DDS at 10 months was the dependent variable, treatment group was the independent variable, and baseline DDS was a covariate. Power calculations were based on effect sizes for the DDS in similar trial that revealed small-to-medium effect sizes. Our goal was to include 130 patients in each arm. The randomized samples (n=138 EPIC, n=135 EUC) exceed the required 130 per group; Test type: Superiority; p = .003, proc mixed in SAS (multilevel modeling); Mean Difference (Final Values) = .32

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from 7/13/2015 to 2/9/2018 (from study initiation to study completion).
Arm/Group | Arm 1: Empowering Patients in Chronic Care (EPIC) | Arm 2: Enhanced Usual Care (EUC)
All-Cause Mortality (participants affected / at risk) | 0/140 | 4/140
Serious Adverse Events (participants affected / at risk) | 0/140 | 0/140
Other Adverse Events (participants affected / at risk) | 0/140 | 0/140

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-17): https://cdn.clinicaltrials.gov/large-docs/85/NCT01876485/Prot_SAP_000.pdf